CLINICAL TRIAL: NCT01710124
Title: Buy 1 Get 1: Role of Grocery Coupons in Promoting Obesogenic Home Food
Brief Title: Buy 1 Get 1: Role of Grocery Coupons in Promoting Obesogenic Home Food Environments and Eating Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 816224
Record Dates: First submitted 2012-10-09; First posted 2012-10-18 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: grocery purchases; financial incentives; obesogenic home food environment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incentive (Experimental): Subjects in this group will receive financial incentives for using grocery coupons to purchase healthy foods.
  Interventions: Other: Financial incentives
- No incentive (No Intervention): Subjects in this group will receive no financial incentives.

INTERVENTIONS:
Other: Financial incentives
  Arms: Incentive

SUMMARY:
The prevalence of overweight and obesity among older adults has reached an all-time high, which puts this age group at high risk for associated comorbidities such as type 2 diabetes, cardiovascular disease, and certain forms of cancer. Confronted with declining incomes and economic uncertainty, many middle-aged and older Americans tried to save on their food purchases during the 2007-2009 recession. Grocery coupons, available through newspapers, mail, and increasingly online, are one of several promotional tools that supermarkets and warehouse clubs use to promote sales. It is estimated that nationally 27% of households are frequent grocery coupon users who shop at a variety of retailers. Despite the increasing popularity of grocery coupons, little is known about the extent to which they may promote obesogenic home food environments and eating behaviors. Many coupons advertise the purchase of large quantities of prepackaged and processed foods and often reward shoppers by adding 'free' products if they purchase certain quantities. Availability and easy accessibility of large portions of energy dense foods in the home has been shown to promote increased intake. The proposed study seeks to examine the effects of frequent grocery coupon usage on dietary intake, weight status, and home food availability among middle-aged and older adults. A second aim of this study is to test, in a randomized-controlled trial, the effects of incentivizing grocery coupon use for the purchase of healthy foods on 3-month changes in dietary intake, body mass index/waist circumference, home food availability, and grocery coupon use among frequent coupon users and non-coupon users.

ELIGIBILITY:
Inclusion Criteria:

* 40 - 70 years of age
* frequent grocery coupon users
* non-coupon users

Exclusion Criteria:

* dieting
* medication use or medical conditions known to affect food intake and weight

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Dietary intake | Change from baseline to month 3 (end of intervention)
Body mass index | Change from baseline to month 3 (end of intervention)
Waist circumference | Change from baseline to month 3 (end of intervention)

SECONDARY OUTCOMES:
Number of healthy and less healthy foods in the home | Change from baseline to month 3 (end of intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States